CLINICAL TRIAL: NCT03425890
Title: The Effect of the Self-empowered Upper Limb Repetitive Engagement (SURE) Program on Upper Limb Recovery Compared With Education in People With Stroke Undergoing Inpatient Rehabilitation
Brief Title: Effect of Self-empowered Upper Limb Repetitive Engagement (SURE) Program on Upper Limb Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National University of Singapore (Other); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Chin Lay Fong, Principal Physiotherapist, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/00600
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: Upper Limb; Self-exercise
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomised Blinded Controlled Pilot Trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to which group the participants are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SURE Program Group (Experimental): The intervention group will receive a SURE program booklet and will perform individualized daily self-exercise and functional use of the arm and hand on their own outside of therapy for 60 minutes/day, 6 days/week for 4 weeks. These self-exercises and upper limb functional use will be performed in addition to usual care. Three SURE program booklets have been developed which relate to the affected upper limb motor capability using individual Fugl Meyer (ULFM) score. Each SURE program booklet consists of warm-up exercises, strengthening exercises and motor tasks. The SURE program booklet also includes selected functional motor tasks to be performed by the participants using their affected upper limb. The performance of the exercises and functional motor tasks will be reviewed three times per week for the first 2 weeks, two times for the third week and one time for the fourth week of intervention period.
  Interventions: Behavioral: SURE program
- Education Group (Experimental): The control group will receive an education booklet with 10 modules. The education booklet will contain information on stroke, recovery and management strategies after stroke. Participants are to complete 2-3 modules per week and answer 1-2 simple questions after each module. Each module including answering questions takes approximately 5-10 minutes to complete. CPI will review the information with the participants 3 times per week for the first 2 weeks, two times for the third week and one time for the fourth week of intervention period.The participants in the control group will continue with their usual care in the hospital.
  Interventions: Behavioral: SURE program

INTERVENTIONS:
Behavioral: SURE program — SURE program is a self-exercise program which aims to empower people with stroke and their caregivers to increase early UL practice outside therapy

SUMMARY:
The aim of this study is to investigate the effect of SURE program on UL recovery during first few weeks post-stroke. A randomised blinded controlled pilot trial will be conducted. Twenty people with stroke will be randomly allocated to 4-weeks of SURE program or education program. This is to perform on top of their usual care. To determine the clinical benefit, all participants will be assessed pre-, 2 weeks during the training, post-training, 1-month and 3-month follow-up using a range of impairment and activity measures. To determine the cortical activation (fMRI), structural (FLAIR and DTI) and functional (resting state fcMRI) connectivity of cortical motor regions, all participants will undergo a 3T MRI pre-, post- and post-3 months after training.

DETAILED DESCRIPTION:
Background:

UL recovery after stroke has been found to be limited. Efforts should be channelled into rehabilitation to improve UL recovery after stroke. First 4-weeks post-stroke is the period when neuroplasticity unfolds and when most rehabilitation occurs. This critical time window should be capitalized to interact with spontaneous biological recovery to facilitate UL recovery. There is growing evidence that shows that early increased UL practice after stroke improves the recovery of upper limb function. However, it has also been found that the level of early UL practice and use during early post-stroke is low. SURE program is a self-exercise program which aims to empower people with stroke and their caregivers to increase early UL practice outside therapy.

Aim:

To investigate the effect of SURE program on UL recovery during first few weeks post-stroke.

Method:

A randomised blinded controlled pilot trial will be conducted. Twenty people with stroke will be randomly allocated to 4-weeks of SURE program or education program.

Intervention Group- SURE Program The intervention group will receive a SURE program booklet and will perform individualized daily self-exercise and functional use of the arm and hand on their own outside of therapy for 60 minutes/day, 6 days/week for 4 weeks. These self-exercises and upper limb functional use will be performed in addition to usual care. Three SURE program booklets have been developed which relate to the affected upper limb motor capability using individual Fugl Meyer (ULFM) score. Each SURE program booklet consists of warm-up exercises, strengthening exercises and motor tasks. The SURE program booklet also includes selected functional motor tasks to be performed by the participants using their affected upper limb. The performance of the exercises and functional motor tasks will be reviewed three times per week for the first 2 weeks, two times for the third week and one time for the fourth week of intervention period.

Control Group- Education The control group will receive an education booklet with 10 modules. The education booklet will contain information on stroke, recovery and management strategies after stroke. Participants are to complete 2-3 modules per week and answer 1-2 simple questions after each module. Each module including answering questions takes approximately 5-10 minutes to complete. CPI will review the information with the participants 3 times per week for the first 2 weeks, two times for the third week and one time for the fourth week of intervention period.The participants in the control group will continue with their usual care in the hospital.

To determine the clinical benefit, all participants will be assessed pre-, 2 weeks during the training, post-training, 1-month and 3-month follow-up using a range of impairment and activity measures. To determine the cortical activation (fMRI), structural (FLAIR and DTI) and functional (resting state fcMRI) connectivity of cortical motor regions, all participants will undergo a 3T MRI pre-, post- and post-3 months after training.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of first-ever stroke occurring less than 21 days ago
2. Positive motor evoked potential on affected hand extensor carpi radialis during Transcranial Magnetic Stimulation (TMS) investigation
3. Clinically moderate to severe UL paresis (ULFM score of less than or equal to 50)
4. Montreal Cognitive Assessment>= 19

Exclusion Criteria:

1. Prior history of central nervous system disorders e.g. Parkinsonism, Spinal Cord Injury, previous stroke
2. Structural brain lesions e.g. brain tumors
3. Medical history of psychiatric disturbance e.g. schizophrenia
4. Bilateral stroke
5. Cardiac disease that limit function by exertional dyspnoea, angina or severe fatigue (defined by physicians and treating therapists)
6. Hemiplegic shoulder pain VAS >5/10
7. Existing peripheral nerve or orthopaedic conditions that interfere with affected UL movement e.g. frozen shoulder, peripheral nerve damage to UL
8. Severe aphasia, neglect, agitation, or depression (defined by physicians and treating therapists) that can limit participation
9. Any contraindications to MRI and TMS.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change of Upper Limb Fugl Meyer Scale (ULFM) | Change from pre training to immediate post training
  Change of Upper Limb Motor Impairment

SECONDARY OUTCOMES:
Change of Upper Limb Fugl Meyer Scale (ULFM) | Change from pre training to 2 weeks into training
  Change of Upper Limb Motor Impairment
Change of Upper Limb Fugl Meyer Scale (ULFM) | Change from 2 weeks into training to immediate post-training
  Change of Upper Limb Motor Impairment
Change of Upper Limb Fugl Meyer Scale (ULFM) | Change from immediate post training to 1-month post-training
  Change of Upper Limb Motor Impairment
Change of Upper Limb Fugl Meyer Scale (ULFM) | Change from 1-month post-training to 3 month post-training
  Change of Upper Limb Motor Impairment
Change of Action Research Arm Test (ARAT) | Change from pre training to 2 weeks into training
  Change of Upper Limb Functional Outcome
Change of Action Research Arm Test (ARAT) | Change from 2 weeks into training to immediate post training
  Change of Upper Limb Functional Outcome
Change of Action Research Arm Test (ARAT) | Change from immediate post training to 1-month post training
  Change of Upper Limb Functional Outcome
Change of Action Research Arm Test (ARAT) | Change from 1-month post training to 3-month post training
  Change of Upper Limb Functional Outcome
Rating of Everyday Arm-Use in the Community and Home (REACH) | Measure at 1-month post training
  Measure real-world use of the arm in everyday tasks
Rating of Everyday Arm-Use in the Community and Home (REACH) | Measure at 3-month post training
  Measure real-world use of the arm in everyday tasks
Stanford Fatigue Visual Numeric Scale (FVNS) | Measure at pre training
  Measure Fatigue Level from 0 point (minimum) to 10 points (maximum) (the higher the score, the more fatigue the participant experience)
Stanford Fatigue Visual Numeric Scale (FVNS) | Measure at 2 weeks into training
  Measure Fatigue Level from 0 point (minimum) to 10 points (maximum) (the higher the score, the more fatigue the participant experience)
Stanford Fatigue Visual Numeric Scale (FVNS) | Measure immediate post training
  Measure Fatigue Level from 0 point (minimum) to 10 points (maximum) (the higher the score, the more fatigue the participant experience)
Visual Analogue Scale (VAS) | Measure at pre training
  Measure Affected UL Pain from 0 point (minimum) to 10 points (maximum) (the higher the score, the more pain the participant experience)
Visual Analogue Scale (VAS) | Measure at 2 weeks into training
  Measure Affected UL Pain from 0 point (minimum) to 10 points (maximum) (the higher the score, the more pain the participant experience)
Visual Analogue Scale (VAS) | Measure at immediate post training
  Measure Affected UL Pain from 0 point (minimum) to 10 points (maximum) (the higher the score, the more pain the participant experience)
Modified Ashworth Scale (MAS) | Measure at pre training
  Measure tone of Affected UL biceps from 0- point (minimum) to 4 points (maximum) (the higher the score, the higher the muscle tone)
Modified Ashworth Scale (MAS) | Measure at 2 weeks into training
  Measure tone of Affected UL biceps from 0- point (minimum) to 4 points (maximum) (the higher the score, the higher the muscle tone)
Modified Ashworth Scale (MAS) | Measure at immediate post training
  Measure tone of Affected UL biceps from 0- point (minimum) to 4 points (maximum) (the higher the score, the higher the muscle tone)
Duration of Affected Upper Limb activity in hours | Measure at 1 week into training
  Measure Duration of Affected Upper Limb activity in hours using Actigraph GT3X-BT wrist accelerometer
Duration of Affected Upper Limb activity in hours | Measure at 2 weeks into training
  Measure Duration of Affected Upper Limb activity in hours using Actigraph GT3X-BT wrist accelerometer
Duration of Affected Upper Limb activity in hours | Measure at 3 weeks into training
  Measure Duration of Affected Upper Limb activity in hours using Actigraph GT3X-BT wrist accelerometer
Duration of Affected Upper Limb activity in hours | Measure at 4 weeks 4 into training
  Measure Duration of Affected Upper Limb activity in hours using Actigraph GT3X-BT wrist accelerometer
Bilateral Motor Cortex Brain Activation | Measure at pre training
  Measuring bilateral motor cortex cortical activation using functional Magnetic Resonance Imaging using a 3T MRI
Bilateral Motor Cortex Brain Activation | Measure at immediate post training
  Measuring bilateral motor cortex cortical activation using functional Magnetic Resonance Imaging using a 3T MRI
Bilateral Motor Cortex Brain Activation | Measure at 3-month post training
  Measuring bilateral motor cortex cortical activation using functional Magnetic Resonance Imaging using a 3T MRI

CONTACTS AND LOCATIONS:
Overall Officials: Lay Fong Chin, Masters, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital Rehabilitation Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participants data to other researchers

DOCUMENTS (1):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03425890/Prot_000.pdf